CLINICAL TRIAL: NCT02431962
Title: Alberta Lung Cancer Screening Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Principal Investigator, Dr. Alain Tremblay, Professor, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10007170
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Lung Neoplasms; Respiratory Tract Neoplasms
Keywords: Lung Cancer; Screening; Computed Tomography
MeSH Terms: conditions — Lung Neoplasms; Respiratory Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Screening arm (Experimental): Annual low dose screening chest CT scan x 3.
  Interventions: Procedure: Computed Tomography
- Smoking cessation counseling (Experimental): Active smokers randomized to this arm will be contacted by a trained smoking cessation counselor and offered cessation support and advice.
  Interventions: Behavioral: Active smokers - Smoking cessation arm
- Smoking cessation control (Active Comparator): Active smokers randomized to this arm will receive general information on available smoking cessation resources.
  Interventions: Behavioral: Active smokers - Control arm

INTERVENTIONS:
Procedure: Computed Tomography — Low dose chest CT screening annually x 3
  Arms: Screening arm
Behavioral: Active smokers - Smoking cessation arm — Phone based smoking cessation counseling
  Arms: Smoking cessation counseling
Behavioral: Active smokers - Control arm — Subjects will be provided with general information on available smoking cessation resources
  Arms: Smoking cessation control

SUMMARY:
Lung cancer is the leading cause of cancer death in North America and in the world. The vast majority of lung cancers are associated with cigarette smoking. Unfortunately, the majority of lung cancers are detected at an advanced stage when they have a very poor prognosis. A substantial amount of data has been reported on low-dose computed tomography (LDCT) screening. Yet endorsement of lung cancer screening has not been universal because of outstanding concerns which need to be addressed. Our study will aim to screen at risk Albertans for lung cancer with LDCT scan at baseline, year 1 and year 2 while attempting to fill some knowledge gaps on this topic.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in North America and in the world. The vast majority of lung cancers are associated with cigarette smoking. Lung cancer incidence and mortality rates are similar because lung cancer is a highly fatal disease. Unfortunately, the majority of lung cancers are detected at an advanced stage when they have a very poor prognosis. A substantial amount of data has been reported on low-dose computed tomography (LDCT) screening. The results of the National Lung Screening Trial (NLST) showed a 20% reduction in mortality from lung cancer with LDCT screening in addition to a 6.7% decrease in all-cause mortality, the first ever screening intervention to demonstrate an improvement in this latter outcome. Yet endorsement of lung cancer screening has not been universal. Although the NLST results are encouraging, more investigation is needed.

The objectives of this study are to prospectively compare the performance of a lung cancer risk prediction model (RPM) vs. NLST criteria to inform optimal inclusion criteria for a clinical screening program; to prospectively compare a novel screening based nodule malignancy probability calculation which has been developed in the Pan-Canadian Early Detection of Lung Cancer study vs. NLST criteria; to complete a randomized controlled trial as a substudy comparing an intensive tobacco cessation counseling program to a usual care arm for subjects with ongoing tobacco use; to perform a cost analysis evaluating the incremental costs associated with LDCT screening for lung cancer compared to no screening; to determine the average cost associated with incidental findings, false positive findings and lung cancers found during the screening period; and to compare cost implications of both screening enrollment criteria.

The backbone of this research project will be the screening of at risk individuals for lung cancer with LDCT scan. Eight hundred at risk Albertans will be screened at baseline, year 1 and year 2. Additional clinical LDCT or other investigations may result from findings on the study CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 55 and 80 with a risk prediction model (RPM) ≥1.5% (≥ 1.5% risk of lung cancer over 6 years) OR NLST criteria (age 55-74; ≥ 30 pack-year smoking history; ongoing smoking or quit within 15 years).
* Ability to provide informed consent and participate in study procedures.

Exclusion Criteria:

* Any medical condition, such as severe heart disease (e.g. unstable angina, chronic congestive heart failure), severe lung disease or lung disease requiring supplemental oxygen that in the opinion of the physician unlikely to benefit from screening due to shortened life-expectancy from the co-morbidities or inability to tolerate diagnosis and treatment of a screen detected abnormality. European Cooperative Oncology Group performance status > 2.
* History of lung cancer.
* Have had other cancer or treatment for cancer within the past 5 years with the exception of the following cancers: non-melanomatous skin cancer, localized prostate cancer, carcinoma in situ (CIS) of the cervix, or superficial bladder cancer. Treatment of the exceptions must have ended > 6 months before registration into this study.
* Pregnancy.
* Hemoptysis in past 12 months.
* Unexplained weight loss >15 pounds / 7kg in past 12 months.
* Unwilling to have a LDCT of chest.
* Unwilling to sign a consent.
* Have had a CT scan of the chest in the last 2 years.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of screening enrollment criteria (Risk prediction model (RPM) vs. NLST criteria) | 5 years
  The proportion of individuals selected by RPM or NLST will be calculated as the number of subjects qualifying and consenting to the screening intervention / total number of subjects enrolled with either criteria. Superiority of the risk prediction model over NLST criteria will be considered established if it identifies at least as many cases of lung cancer as the NLST while sampling fewer individuals.
Randomized trial of smoking cessation intervention in screened individuals (smoking status [smoking rates assessed via questionnaire and abstinence confirmed by saliva nicotine or exhaled carbon minoxide]) | 3 years
  The primary study endpoint will be an assessment of smoking status at 12 months following randomization. Smoking rates will be assessed via phone questionnaire and abstinence confirmed by saliva nicotine test or exhaled carbon monoxide in subjects using nicotine replacement therapies (to avoid false positive nicotine test).

SECONDARY OUTCOMES:
Evaluation of nodule risk calculator | 3 years
  We will prospectively validate a nodule risk calculator by comparing the proportion of baseline CT examinations reported as positive by the calculator vs. NLST criteria on a per subject basis
Health Economics Analysis (healthcare payer and all direct health-care related cost) | 4 years
  Costs will be estimated for the cohort of individuals who enroll in the screening program and consent to receive a LDCT scan. Costs will also be estimated for a group of individuals who are eligible for the screening program however do not undergo screening. We will include costs for all relevant health care categories for a 2 year period from the date of risk stratification. The perspective of the analysis will be that of the healthcare payer and all direct health-care related costs would be captured and reported in Canadian dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Tremblay, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Derived] Tremblay A, Taghizadeh N, MacEachern P, Burrowes P, Graham AJ, Lam SC, Yang H, Koetzler R, Tammemagi MC, Taylor K, Bedard ELR. Two-Year Follow-Up of a Randomized Controlled Study of Integrated Smoking Cessation in a Lung Cancer Screening Program. JTO Clin Res Rep. 2020 Sep 15;2(2):100097. doi: 10.1016/j.jtocrr.2020.100097. eCollection 2021 Feb. PMID 34589978
- [Derived] Tremblay A, Taghizadeh N, Huang J, Kasowski D, MacEachern P, Burrowes P, Graham AJ, Dickinson JA, Lam SC, Yang H, Koetzler R, Tammemagi M, Taylor K, Bedard ELR. A Randomized Controlled Study of Integrated Smoking Cessation in a Lung Cancer Screening Program. J Thorac Oncol. 2019 Sep;14(9):1528-1537. doi: 10.1016/j.jtho.2019.04.024. Epub 2019 May 8. PMID 31077790